CLINICAL TRIAL: NCT06693219
Title: Accuracy of Ultrasonography in Confirming Correct Positioning of Nasogastric Tube in the Intensive Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-00036
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Nasogastric Tube Placement; Accuracy; Ultrasonography; Critical Care, Intensive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (Experimental)
  Interventions: Diagnostic Test: ultrasonography to confirm the correct placement of a nasogastric tube in the stomach

INTERVENTIONS:
Diagnostic Test: ultrasonography to confirm the correct placement of a nasogastric tube in the stomach — The sonographic examination consisted of three parts: neck scan, epigastric scan, and injection test using a mixture of 25 mL NaCl 0.9% and 25 mL room air through the nasogastric tube to detect dynamic fogging

SUMMARY:
The goal of the study was to test whether a sonographic examination instead of an X-ray allows the position of a tube in the stomach to be checked.

Participants were patients admitted at an intensive care unit who required a nasogastric tube for several reasons (for example nutrition). After obtaining an informed consent from the patient or the family, the researchers checked the position of the tube with ultrasound and compared it with the gold standard, which is radiography. Data analysis allowed the concordance between the two tests to be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* an already inserted nasogastric tube or required nasogastric tube insertion
* no contraindication for chest or abdominal X-ray
* no contraindication for neck and upper abdominal ultrasonography

Exclusion Criteria:

* pregnancy
* basal skull fractures
* facial fractures
* previous or recent surgery of the neck, esophagus or stomach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of ultrasonography in determining correct nasogastric tube placement in the stomach | Through study completion (enrollment of approximately 180 patients)
  In order to assess its diagnostic accuracy (sensitivity, specificity, negative predictive value, positive predictive value) we compared the index test (ultrasonography) against the reference standard (X-ray)

CONTACTS AND LOCATIONS:
Locations (1):
- Medicina Intensiva, Ente ospedaliero cantonale, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No